CLINICAL TRIAL: NCT02121353
Title: A Pilot Phase 1/2, Double Blind, Parallel Group, Controlled Study of the Safety, Tolerability and Preliminary Efficacy Evaluation of Intravitreally Administered Pfenex Ranibizumab Biosimilar Versus Lucentis for the Treatment of Neovascular AMD
Brief Title: Safety Study of PF582 Versus Lucentis in Patients With Age Related Macular Degeneration
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfenex, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PF582-CLIN-001
Record Dates: First submitted 2014-04-17; First posted 2014-04-23 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Age Related Macular Degeneration (AMD)
Keywords: Age related macular degeneration; AMD; Wet AMD; Eye conditions; CFT; OCT; CNV; FA; Ocular; Eye; Disorder of the eye
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PF582 (Experimental): PF582 is provided as single use vials and will be administered by intra-vitreal injection on Day 1, 28 and 56.
  Interventions: Drug: PF582
- Lucentis (Active Comparator): Lucentis® is provided as single use vials and will be administered by intra-vitreal injection on Day 1, 28 and 56.
  Interventions: Drug: Lucentis

INTERVENTIONS:
Drug: Lucentis — Single-use 2 mL vial designed to deliver 0.05 mL of 10 mg/mL ranibizumab solution. Excipients: Alpha, alpha-trehalose dihydrate; histidine hydrochloride, monohydrate; histidine; polysorbate 20; water for injections Route of Administration: Intra-vitreal
  Other Names: ranibizumab
  Arms: Lucentis
Drug: PF582 — Single-use 2 mL vial designed to deliver 0.05 mL of 10 mg/mL ranibizumab solution. Excipients: Alpha, alpha-trehalose dihydrate; histidine hydrochloride, monohydrate; histidine; polysorbate 20; water for injections Route of Administration: Intra-vitreal
  Other Names: ranibizumab
  Arms: PF582

SUMMARY:
The aim of this study is to test if PF582 (ranibizumab) is safe and similar to Lucentis (ranibizumab). Participants will have a screening visit to check for eligibility. Eligible participants will receive either PF582 or Lucentis, by injection into one eye on study Day 1, 28 and 56. Visits will be conducted on Day 2, 7, 14 80 and at 6 and 12 months. During the study participants will undergo the following procedures: height, weight and vital signs (blood pressure, pulse, temperature, breathing rate) measurement; medical and surgical history and concomitant medications; adverse event monitoring; physical examinations; eye tests (reading chart, measurement of retinal thickness [via pictures of the retina] and examination of the eye's blood vessels, via pictures taken following injection of a dye into the arm), blood collection and a urine pregnancy test, where applicable.

DETAILED DESCRIPTION:
To evaluate the safety and tolerability of PF582, compared to that of Lucentis (registered trademark) in patients with neovascular AMD. This will be done by assessment of vital signs, physical examination, laboratory blood tests and adverse events. Possible adverse events include: eye irritation/discomfort, redness/itching eye, eye dryness, abnormal sensation in eye; lens clouding; pain/irritation at injection site; increased tear production; 'floaters'; sore throat, nasal congestion, headache, joint pain, flu, fatigue, breathlessness, dizziness, pale skin, anxiety, cough, nausea and allergic reactions.

Because PF582 is very similar to Lucentis it is expected to have similar adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥50 years
* Presence in the study eye (one eye per patient) of previously untreated active subfoveal CNV due to AMD, with presence of leakage, as seen on FA, and of fluid, as seen on spectral-domain OCT, located either within or below the retina, or below the retinal pigment epithelium
* Visual acuity between 20/25 and 20/320 being measured using the Early treatment diabetic retinopathy study (ETDRS) protocol1 (chart at 4 meters) before pupil dilation.
* Neovascularization, fluid, or haemorrhage under the fovea.
* Fibrosis < 50% of total lesion area
* At least 1 drusen (>63μm) in either eye or late AMD in fellow eye.
* Female subjects must be of non-childbearing potential, meeting at least one of the following criteria:
* Amenorrheal for 12 months (Menopause confirmed by FSH and LH levels as defined by the established reference ranges), or taking oral contraception for at least 3 months, or surgically sterile for at least the past 3 months, or Receiving a stable dose of implanted or injectable contraceptive for at least 3 months

Exclusion Criteria:

* Previous treatment for CNV in study eye, including antivascular endothelial growth factor(VEGF) medication
* Other progressive retinal disease in the study eye, or the non-study eye, likely to compromise Visual Acuity assessment.
* Contraindications to injections with Lucentis®
* Sub-retineal Haemorrhage > 50% of lesion
* Fibrosis or retrofoveolar atrophy
* History of retrofoveolar laser photocoagulation
* Previous Lucentis® treatment
* Any other treatment (photocoagulation, phototherapy, radiotherapy, surgery, thermotherapy) in the last 3 months
* Aphaky, vitrectomy
* Active or suspected ocular or periocular infection
* Active intraocular inflammation
* Active systemic infection
* History of stroke or congestive heart failure
* Any other clinical significant illness or abnormalities that would compromise the safety of the participant
* Inability to comply with study or follow up procedures

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of PF582 | Up to 12 months
  To evaluate the safety and tolerability of PF582, compared to that of Lucentis (registered trademark) in patients with neovascular AMD. This will be done by assessment of vital signs, physical examination, laboratory blood tests and adverse events. Possible adverse events include: eye irritation/discomfort, redness/itching eye, eye dryness, abnormal sensation in eye; lens clouding; pain/irritation at injection site; increased tear production; 'floaters'; sore throat, nasal congestion, headache, joint pain, flu, fatigue, breathlessness, dizziness, pale skin, anxiety, cough, nausea and allergic reactions. Because PF582 is very similar to Lucentis it is expected to have similar adverse effects.

SECONDARY OUTCOMES:
To demonstrate the biosimiliarity between PF582 and Lucentis based on PK | up to 12 months
  To demonstrate the biosimiliarity between PF582 and the reference compound (Lucentis) based on pharmacokinetics (PK). This will be done by collection and analysis of PK blood samples.
To demonstrate biosimilarity between PF582 and reference compound (Lucentis) | 12 months
  Preliminary analysis of efficacy, as evaluated by mean change in visual acuity between baseline and Day 80 assessment, and proportion of patients with a change in visual acuity of 15 letters or more

OTHER OUTCOMES:
To demonstrate the biosimiliarity between PF582 and the reference compound (Lucentis), based on pharmacodynamics (PD) parameters. | Up to 12 months
  To demonstrate the biosimiliarity between PF582 and the reference compound (Lucentis), based on pharmacodynamics (PD) parameters. This will be assessed by measuring retinal thickness or central foveal thickness (CFT), assessed by optical coherence tomography (OCT)), Leakage from choroidal neovascularization (CNV) assessed by fluorescein angiography (FA).

CONTACTS AND LOCATIONS:
Overall Officials: Philip Polkinghorne, MD, Principal Investigator; Hubert C Chen, MD, Study Director — Pfenex, Inc
Locations (2):
- New Zealand (2):
  - Eye Institute, Remuera, Auckland
  - Auckland Eye 8 St Marks Road Remuera Auckland 1050, Auckland